CLINICAL TRIAL: NCT05754333
Title: A Phase 3, Multicenter, Prospective, Randomized, Open-label Study for Intraoperative Ureter(s) Visualization When Using ASP5354 With Near Infrared Fluorescence (NIR-F) Imaging in Participants Undergoing Minimally Invasive and Open Abdominopelvic Surgeries
Brief Title: A Study to Find Out if ASP5354 Can Clearly Help Show the Ureter During Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5354-CL-0301
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Intraoperative Ureter Visualization; Abdominolpelvic Surgery
Keywords: ASP5354; pudexacianinium chloride; Iatrogenic ureteral injury; Abdominopelvic surgery; Near infrared fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Adult (Normal/Mild): White Light/near-infrared fluorescence (Experimental): Adults participants with with normal renal function or mild renal impairment received a single IV 3 mg dose (3 vials of 1 mg) of pudexacianinium chloride administered approximately 30 (± 15) min before ureter visualization, on day 1. WL and NIR-F were used to recognize/identify the ureter.
  Interventions: Drug: pudexacianinium chloride
- Adult (Normal/Mild): White Light only (Experimental): Adults participants with normal renal function or mild renal impairment received a single IV 3 mg dose (3 vials of 1 mg) of pudexacianinium chloride approximately 30 (± 15) min before the ureter visualization, on day 1. WL was used to recognize/identify the ureter.
  Interventions: Drug: pudexacianinium chloride
- Adult (Moderate): White Light/near-infrared fluorescence (Experimental): Adults participants with moderate renal impairment received a single IV 3 mg dose (3 vial of 1 mg) of pudexacianinium chloride approximately 30 (± 15) min before ureter visualization, on day 1. WL and NIR-F were used to recognize/identify the ureter.
  Interventions: Drug: pudexacianinium chloride
- Adolescent (Normal/Mild): White Light/near-infrared fluorescence (Experimental): Adolescents participants with normal renal function or mild renal impairment renal impairment received a single IV 3 mg dose (3 vials of 1 mg) of pudexacianinium chloride approximately 30 (± 15) min before ureter visualization, on day 1. WL and NIR-F were used to recognize/identify the ureter.
  Interventions: Drug: pudexacianinium chloride

INTERVENTIONS:
Drug: pudexacianinium chloride — Intravenous
  Other Names: ASP5354

SUMMARY:
The ureter was the tube that carries urine from the kidneys to the bladder. It was difficult for surgeons to see the ureter during abdominal surgery. This could lead to injuring the ureter which, although rare, could be serious. This study was about a potential new medical dye, called ASP5354. This dye was injected into the person at the start of surgery and was detected in the ureter. This was done by an imaging machine which had an option called near infrared fluorescence, or NIR-F. Together they showed live images of specific parts of the body. In this study, ASP5354 was used with an imaging machine with a NIR-F option to show live images of the ureter during surgery. People with kidneys that work properly and those with kidney problems could take part. The main aim of the study was to find out how clearly the ureter could be seen with ASP5354 during surgery in adults whose kidneys work properly or who have mild kidney problems. To do this, the surgeons injected ASP5354 into the person having surgery. Then, the surgeons compared images of the ureter with an imaging machine using normal white light and with the NIR-F option. Imaging using normal white light was the standard way surgeons see the ureter during surgery. People 12 years or older who were going to have certain abdominal surgeries could take part. Everyone taking part received ASP5354 during surgery, but how the imaging was done depended on which group they are in. Before surgery, the adults taking part whose kidneys work properly or who have mild kidney problems were assigned into 1 of 2 groups by chance alone. Images of the ureter were checked in 1 group using normal white light and the other group using normal white light and NIR-F. People 18 years and older with more severe kidney problems and all people under 18 years old were not be assigned to 1 of 2 groups: all images of the ureter were checked using normal white light and NIR-F. At the start of surgery, the surgeon injected ASP5354 into the person having surgery, then started recording a video. Then, after 30 minutes, the surgeon recorded how well the ureter could be seen. This was done by either using normal white light, or normal white light and NIR-F, depending which group each person having surgery was assigned to. For the group to be checked with normal white light and NIR-F, the surgeon did this every 30 minutes until the end of surgery. For the group to be checked with normal white light only, the surgeon did this after the first 30 minutes. During the study, people visited the study hospital 3 times. The first visit was to check if they can take part in the study. People were asked about their medical history, have had a medical examination, and their vital signs checked (blood pressure and pulse rate). Also, they had some blood and urine tests. For women and girls this may included a pregnancy test. People had their surgery at the second visit. This was within 28 days of their first visit. This included having some blood and urine tests before, during, and after surgery. Also, they had a medical examination, an electrocardiogram (ECG) to check their heart rhythm, and had their vital signs checked. After surgery, people returned to the clinic 15 days later for a final check-up. They were asked if they have had any medical problems. Also, they had a medical examination, had their vital signs checked, and had some blood and urine tests.

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled to undergo minimally invasive or open abdominopelvic surgery that may require ureter(s) identification.
* Participant has normal renal function or has varying degrees of chronic kidney disease as defined by the National Kidney Foundation and calculated by individual eGFR using the modification of diet in renal disease (MDRD) formula for adults or the Schwartz formula for adolescents at the screening visit.

  * Adult normal/mild eGFR cohort: eGFR ≥ 60 mL/min
  * Adult moderate/severe eGFR cohort: eGFR ≥ 15 to < 60 mL/min
  * Adolescent cohort: eGFR ≥ 60 mL/min
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP).
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after study intervention administration.
* Female participant must agree not to breastfeed starting at the administration of ASP5354 through 30 days after ASP5354 administration.
* Female participant must not donate ova starting at the administration of ASP5354 through 30 days after ASP5354 administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception through at least 30 days after ASP5354 administration.
* Male participant must not donate sperm starting at the administration of ASP5354 through 30 days after ASP5354 administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy from the start of ASP5354 administration through 30 days after ASP5354 administration.
* Participant (and/or participant's parent or legal guardian) agrees not to participate in another interventional study involving unapproved study medication while participating in the present study.

Exclusion Criteria:

* Participant has any physical or psychiatric condition which makes the participant unsuitable for study participation.
* Participant is anticipated to require ureteral stenting during surgery.
* Participant has an active urinary tract infection requiring antibiotic therapy.
* Participant has moderate to severe cardiac disease that limits daily functioning (New York Heart Association Class III to IV) or other medical conditions that would impact safety or study compliance.
* Participant has any clinically relevant laboratory abnormality that could contraindicate surgery.
* Participant with body weight < 30 kilogram (kg).
* Participant has a known or suspected hypersensitivity to ASP5354, indocyanine green (ICG) or any components of the formulation used.
* Participant has had previous exposure to ASP5354.
* Participant has been administered ICG or other near-infrared fluorescent (NIR-F) imaging agents within 48 hours prior to ASP5354 administration, with the exception of participants who receive ICG for lymphatic mapping before the surgery.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to randomization.
* Participant is on hemodialysis, hemodiafiltration or peritoneal dialysis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (6):
- United States (6):
  - AdventHealth Orlando, Orlando, Florida
  - Advent Health Tampa, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with normal renal function or mild renal impairment [estimated glomerular filtration rate (eGFR) ≥ 60 mililiter/minute (mL/min)], or adults with moderate or severe renal impairment [eGFR ≥ 15 to < 60 mL/min] and adolescents with normal renal function or mild renal impairment [eGFR ≥ 60 mL/min]) were enrolled in the study. There were no participants enrolled with severe renal impairment.
Pre-assignment Details: Participants who met inclusion criteria and none of the exclusion criteria were enrolled in the study. Randomization was stratified by type of surgery: gynecological abdominopelvic
Groups:
- Adult (Normal/Mild): White Light/Near-infrared Fluorescence: Pudexacianinium (3 milligrams [mg]) was administered as a single intravenous (IV) dose approximately 30 minutes (min) before ureter visualization, on Day 1 in adult participants with normal renal function or mild renal impairment. White Light (WL) and near-infrared fluorescence (NIR-F) were used to recognize/identify the ureter.
- Adult (Normal/Mild): White Light Only: Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult participants with normal renal function or mild renal impairment. WL was used to recognize/identify the ureter.
- Adult (Moderate): White Light/Near-infrared Fluorescence: Pudexacianinium (3mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult participants with moderate renal impairment. WL and NIR-F were used to recognize/identify the ureter.
- Adolescent (Normal/Mild): White Light/Near-infrared Fluorescence: Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adolescent participants with normal renal function or mild renal impairment. WL and NIR-F were used to recognize/identify the ureter.
Period: Overall Study
Arm/Group | Adult (Normal/Mild): White Light/Near-infrared Fluorescence | Adult (Normal/Mild): White Light Only | Adult (Moderate): White Light/Near-infrared Fluorescence | Adolescent (Normal/Mild): White Light/Near-infrared Fluorescence
Started | 72 | 13 | 8 | 14
Participants Did Not Receive Study Drug | 2 | 0 | 0 | 0
Modified Intent-to-Treat (mITT) | 72 | 0 | 8 | 14
Intent-to-Treat (ITT) | 72 | 0 | 0 | 0
Safety Analysis Set (SAF) | 70 | 13 | 8 | 14
Completed | 67 | 12 | 8 | 13
Not Completed | 5 | 1 | 0 | 1
Not completed — Miscellaneous | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: SAF
Groups:
- Adult (Normal/Mild): White Light/Near-infrared Fluorescence: Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult participants with normal renal function or mild renal impairment. WL and NIR-F were used to recognize/identify the ureter.
- Adolescent (Normal/Mild): WL/NIR-F: Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adolescent participants with normal renal function or mild renal impairment. WL and NIR-F were used to recognize/identify the ureter.
- Total: Total of all reporting groups
Arm/Group | Adult (Normal/Mild): White Light/Near-infrared Fluorescence | Adult (Normal/Mild): White Light Only | Adult (Moderate): White Light/Near-infrared Fluorescence | Adolescent (Normal/Mild): WL/NIR-F | Total
Number analyzed (Participants) | 70 | 13 | 8 | 14 | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (15.0) | 52.2 (21.6) | 70.3 (8.6) | 14.4 (1.7) | 49.9 (20.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 10 | 6 | 8 | 72
  Male | 22 | 3 | 2 | 6 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 1 | 2 | 4 | 18
  Not Hispanic or Latino | 57 | 12 | 6 | 10 | 85
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 0 | 1 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 2 | 0 | 1 | 12
  White | 51 | 11 | 7 | 12 | 81
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 0 | 0 | 5
Type of Surgery (Gynecological & Other-Abdominopelvic) [Number; unit: Participants]
  Gynecological | 15 | 2 | 0 | 7 | 24
  Other- Abdominopelvic | 55 | 11 | 8 | 7 | 81

OUTCOME MEASURES:

1. Primary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL and NIR-F at 30 Minutes [Adult (Normal/Mild): WL/NIR-F]
Description: Ureter conspicuity was scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 to 5 where 1= none (not self-evident), 2= poor (somewhat self-evident), 3= sufficient (sufficiently self-evident), 4= good (clearly self-evident), 5= excellent (extremely self-evident). All participants had conspicuity scores from one ureter.
Time Frame: 30 minutes post dose (+/- 15 minutes)
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL): Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult participants with normal renal function or mild renal impairment. WL and NIR-F were used to recognize/identify the ureter. WL was reported for this arm.
- Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F): Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult participants with normal renal function or mild renal impairment. WL and NIR-F were used to recognize/identify the ureter. NIR-F was reported for this arm.
Arm/Group | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 72 | 72
score on a scale | 2.7 (1.5) | 4.3 (1.2)
Statistical Analysis 1: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; p < 0.001, paired t Test; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [1.2 to 1.9], Standard Error of Mean 0.2 — Mean Difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint

2. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F an Average of All Timepoints [Adult (Normal/Mild): WL/NIR-F]
Description: as for outcome 1
Time Frame: WL: 30 minutes (+/- 15 minutes); NIR-F: 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 450, 480 minutes
Population: ITT with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 72 | 72
score on a scale
  30 minutes | 2.7 (1.5) | 4.3 (1.2)
  60 minutes: number analyzed (Participants) | 0 | 50
  60 minutes |  | 4.3 (1.2)
  90 minutes: number analyzed (Participants) | 0 | 45
  90 minutes |  | 4.2 (1.1)
  120 minutes: number analyzed (Participants) | 0 | 33
  120 minutes |  | 4.2 (1.1)
  150 minutes: number analyzed (Participants) | 0 | 23
  150 minutes |  | 3.8 (1.4)
  180 minutes: number analyzed (Participants) | 0 | 17
  180 minutes |  | 3.8 (1.3)
  210 minutes: number analyzed (Participants) | 0 | 9
  210 minutes |  | 3.9 (1.7)
  240 minutes: number analyzed (Participants) | 0 | 3
  240 minutes |  | 4.7 (0.6)
  270 minutes: number analyzed (Participants) | 0 | 4
  270 minutes |  | 4.5 (1.0)
  300 minutes: number analyzed (Participants) | 0 | 2
  300 minutes |  | 5.0 (0.0)
  330 minutes: number analyzed (Participants) | 0 | 1
  330 minutes |  | 4.0 (NA) — Only 1 participant was analyzed hence SD was not evaluable
  450 minutes: number analyzed (Participants) | 0 | 1
  450 minutes |  | 1.0 (NA) — Only 1 participant was analyzed hence SD was not evaluable
  480 minutes: number analyzed (Participants) | 0 | 2
  480 minutes |  | 4.0 (1.4)
Statistical Analysis 1: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; p < 0.001, Sign test; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [1.2 to 1.8], Standard Error of Mean 0.2 — Mean Difference was calculated by averaging over the differences between NIR-F scores at each time point and the 30-min WL score of the index ureter (left or right) for each participant

3. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F at End of Surgery [Adult (Normal/Mild): WL/NIR-F]
Description: as for outcome 1
Time Frame: WL: 30 minute post dose (+/- 15 minutes); NIR-F: End of surgery (Day 1)
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 72 | 72
score on a scale
  30 minutes: number analyzed (Participants) | 72 | 0
  30 minutes | 2.7 (1.5) |
  End of surgery (Day 1): number analyzed (Participants) | 0 | 72
  End of surgery (Day 1) |  | 4.0 (1.3)
Statistical Analysis 1: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; p < 0.001, paired t test; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [1.0 to 1.7], Standard Error of Mean 0.2 — Mean Difference was calculated by averaging over the differences between WL score at 30-min time point and the NIR-F score at the end of surgery across all participants

4. Secondary Outcome: Quantification of Ureter Conspicuity for WL and NIR-F Illumination Modes [Adult (Normal/Mild): WL/NIR-F]
Description: UC was quantified by image analysis when pudexacianinium was present in ureter. Contrast enhancement factor (CEF) was measure of degree to which color contrast (CC) was enhanced in areas in which drug fluorescence signal was present. Images of ureters during surgery were decomposed into red (R), green (G) & blue (B) using Image analysis software. R, G & B video components corresponding to each full color image were exported as 256 shades of gray, ranging from pure black (0) to pure white (255). CC between dye fluorescence in ureter & surrounding tissues was quantified by calculating ratio of signal levels G/(R + B). A higher CEF score=higher (green) contrast in ureter compared to the surrounding tissue. A commensurate ratio value was calculated for signals emanating from tissues surrounding ureter lumen. A comparison of ratio values was expressed as a CEF = (G/(R + B)inside)/(G/(R + B)outside. Overall average data of each time point from first dose up to end of surgery was reported.
Time Frame: From first dose every 30 minutes thereafter up to end of surgery (Day 1)
Population: ITT
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 72 | 72
ratio | 1.08 (0.15) | 2.38 (1.54)

5. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL and NIR-F at 30 Minutes [Adolescent (Normal/Mild): WL/NIR-F]
Description: as for outcome 1
Time Frame: 30 minutes post dose (+/- 15 minutes)
Population: Modified Intent to Treat (mITT): All adolescent participants in the WL/NIR-F arm
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL): Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adolescent participants with normal renal function or mild renal impairment. WL and NIR-F were used to recognize/identify the ureter. Only WL was reported for this arm.
- Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F): Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adolescent participants with normal renal function or mild renal impairment. WL and NIR-F were used to recognize/identify the ureter. Only NIR-F was reported for this arm.
Arm/Group | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 14 | 14
score on a scale | 3.5 (1.5) | 4.4 (1.2)
Statistical Analysis 1: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; Mean Difference (Final Values) = 0.9, Standard Error of Mean 0.3 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint

6. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F an Average of All Timepoints [Adolescent (Normal/Mild): WL/NIR-F]
Description: as for outcome 1
Time Frame: WL: 30 minutes(+/- 15 minutes); NIR-F: 30, 60, 90, 120, 150, 180, 210 minutes
Population: mITT in adolescents with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 14 | 14
score on a scale
  30 minutes | 3.5 (1.5) | 4.4 (1.2)
  60 minutes: number analyzed (Participants) | 0 | 11
  60 minutes |  | 4.5 (0.5)
  90 minutes: number analyzed (Participants) | 0 | 4
  90 minutes |  | 4.5 (0.6)
  120 minutes: number analyzed (Participants) | 0 | 1
  120 minutes |  | 5.0 (NA) — Only 1 participant was analyzed hence SD was not evaluable
  150 minutes: number analyzed (Participants) | 0 | 1
  150 minutes |  | 4.0 (NA) — Only 1 participant was analyzed hence SD was not evaluable
  180 minutes: number analyzed (Participants) | 0 | 1
  180 minutes |  | 4.0 (NA) — Only 1 participant was analyzed hence SD was not evaluable
  210 minutes: number analyzed (Participants) | 0 | 1
  210 minutes |  | 2.0 (NA) — Only 1 participant was analyzed hence SD was not evaluable
Statistical Analysis 1: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; Mean Difference (Final Values) = 1.0, Standard Error of Mean 0.3 — Mean Difference was calculated by averaging over the differences between NIR-F scores at each time point and the 30-min WL score of the ureter of interest (left; right) for each participant

7. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F at End of Surgery [Adolescent (Normal/Mild): WL/NIR-F]
Description: as for outcome 1
Time Frame: WL: 30 minute post dose (+/- 15 minutes); NIR-F: End of surgery (Day 1)
Population: mITT in adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 14 | 14
score on a scale
  30 minutes: number analyzed (Participants) | 14 | 0
  30 minutes | 3.5 (1.5) |
  End of surgery (Day 1): number analyzed (Participants) | 0 | 14
  End of surgery (Day 1) |  | 4.4 (0.9)
Statistical Analysis 1: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; Mean Difference (Final Values) = 0.9, Standard Error of Mean 0.4 — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL and NIR-F at 30 Minutes [Adult (Moderate): WL/NIR-F]
Description: as for outcome 1
Time Frame: 30 minutes post dose (+/- 15 minutes)
Population: mITT in adults with moderate eGFR in the WL/NIR-F arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL): Pudexacianinium (3mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult participants with moderate renal impairment. WL and NIR-F were used to recognize/identify the ureter. Only WL was reported for this arm.
- Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F): Pudexacianinium (3mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult participants with moderate renal impairment. WL and NIR-F were used to recognize/identify the ureter. Only NIR-F was reported for this arm.
Arm/Group | Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) | Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 8 | 8
score on a scale | 1.4 (0.7) | 2.9 (1.1)
Statistical Analysis 1: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; Mean Difference (Final Values) = 1.5, Standard Error of Mean 0.3 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint

9. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F an Average of All Timepoints [Adult (Moderate): WL/NIR-F]
Description: as for outcome 1
Time Frame: WL: 30 minutes(+/- 15 minutes); NIR-F: 30, 60, 90, 120, 150, 180 minutes
Population: mITT in adults with moderate eGFR with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F): Pudexacianinium (3mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult participants with moderate renal impairment. WL and NIR-F were used to recognize/identify the ureter. Only WL was reported for this arm.
Arm/Group | Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) | Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 8 | 8
score on a scale
  30 minutes | 1.4 (0.7) | 2.9 (1.1)
  60 minutes: number analyzed (Participants) | 0 | 5
  60 minutes |  | 4.2 (1.1)
  90 minutes: number analyzed (Participants) | 0 | 5
  90 minutes |  | 3.2 (1.6)
  120 minutes: number analyzed (Participants) | 0 | 5
  120 minutes |  | 3.8 (1.1)
  150 minutes: number analyzed (Participants) | 0 | 3
  150 minutes |  | 2.7 (1.5)
  180 minutes: number analyzed (Participants) | 0 | 1
  180 minutes |  | 2.0 (NA) — Only 1 participant was analyzed hence SD was not evaluable
Statistical Analysis 1: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; Mean Difference (Final Values) = 1.9, Standard Error of Mean 0.2 — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F at End of Surgery [Adult (Moderate): WL/NIR-F]
Description: as for outcome 1
Time Frame: WL: 30 minute post dose (+/- 15 minutes); NIR-F: End of surgery (Day 1)
Population: mITT in adults with moderate eGFR.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) | Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 8 | 8
score on a scale
  30 minutes: number analyzed (Participants) | 8 | 0
  30 minutes | 1.4 (0.7) |
  End of Surgery (Day1): number analyzed (Participants) | 0 | 8
  End of Surgery (Day1) |  | 2.9 (1.5)
Statistical Analysis 1: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; Mean Difference (Final Values) = 1.5, Standard Error of Mean 0.6 — Mean Difference is calculated by averaging over the differences between WL score at 30-min time point and the NIR-F score at the end of surgery across all participants

11. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL and NIR-F at 30 Minutes [All Participants]
Description: as for outcome 1
Time Frame: 30 minutes post dose (+/- 15 minutes)
Population: mITT that included all participants in any cohort in the WL/NIR-F arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: White Light +Near-infrared Fluorescence (Only WL): Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult and adolescent participants with normal renal function or mild or moderate renal impairment. WL and NIR-F were used to recognize/identify the ureter. Only WL was reported for this arm.
- All Participants: White Light +Near-infrared Fluorescence (Only NIR-F): Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult and adolescent participants with normal renal function or mild or moderate renal impairment. WL and NIR-F were used to recognize/identify the ureter. Only NIR-F was reported for this arm.
Arm/Group | All Participants: White Light +Near-infrared Fluorescence (Only WL) | All Participants: White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 94 | 94
score on a scale | 2.7 (1.6) | 4.2 (1.2)
Statistical Analysis 1: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; Mean Difference (Final Values) = 1.4, Standard Error of Mean 0.1 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint

12. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F an Average of All Timepoints [All Participants]
Description: as for outcome 1
Time Frame: WL: 30 minutes(+/- 15 minutes); NIR-F: 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 450, 480 minutes
Population: mITT for all cohorts in WL/NIR-F arm with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants: White Light +Near-infrared Fluorescence (Only WL) | All Participants: White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 94 | 94
score on a scale
  30 minutes | 2.7 (1.6) | 4.2 (1.2)
  60 minutes: number analyzed (Participants) | 0 | 66
  60 minutes |  | 4.3 (1.3)
  90 minutes: number analyzed (Participants) | 0 | 54
  90 minutes |  | 4.1 (1.1)
  120 minutes: number analyzed (Participants) | 0 | 39
  120 minutes |  | 4.2 (1.1)
  150 minutes: number analyzed (Participants) | 0 | 27
  150 minutes |  | 3.7 (1.4)
  180 minutes: number analyzed (Participants) | 0 | 19
  180 minutes |  | 3.7 (1.3)
  210 minutes: number analyzed (Participants) | 0 | 10
  210 minutes |  | 3.7 (1.7)
  240 minutes: number analyzed (Participants) | 0 | 3
  240 minutes |  | 4.7 (0.6)
  270 minutes: number analyzed (Participants) | 0 | 4
  270 minutes |  | 4.5 (1.0)
  300 minutes: number analyzed (Participants) | 0 | 2
  300 minutes |  | 5.0 (0.0)
  330 minutes: number analyzed (Participants) | 0 | 1
  330 minutes |  | 4.0 (NA) — Only 1 participant was analyzed hence SD was not evaluable
  450 minutes: number analyzed (Participants) | 0 | 1
  450 minutes |  | 1.0 (NA) — Only 1 participant was analyzed hence SD was not evaluable
  480 minutes: number analyzed (Participants) | 0 | 2
  480 minutes |  | 4.0 (1.4)
Statistical Analysis 1: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; Mean Difference (Final Values) = 1.4, Standard Error of Mean 0.1 — [estimate comment as in outcome 6, analysis 1]

13. Secondary Outcome: Investigator Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F at End of Surgery [All Participants]
Description: as for outcome 1
Time Frame: WL: 30 minute post dose (+/- 15 minutes); NIR-F: End of surgery (Day 1)
Population: mITT for all cohorts in WL/NIR-F arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants: White Light +Near-infrared Fluorescence (Only WL) | All Participants: White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 94 | 94
score on a scale
  30 minutes: number analyzed (Participants) | 94 | 0
  30 minutes | 2.7 (1.6) |
  End of surgery (Day 1): number analyzed (Participants) | 0 | 94
  End of surgery (Day 1) |  | 4.0 (1.3)
Statistical Analysis 1: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; Mean Difference (Final Values) = 1.3, Standard Error of Mean 0.2 — [estimate comment as in outcome 3, analysis 1]

14. Secondary Outcome: Percentage of Participants (POP) With an Average Index Ureter Conspicuity Under NIR-F at Least 1, 2, 3 or 4 Point Higher Than the Average Index Ureter Conspicuity Under WL Over All Time Points [All Participants]
Description: Ureter conspicuity was scored individually for each illumination mode using a 5-Point Likert Scale, ranging from 1 to 5 where 1= none (not self-evident), 2= poor (somewhat self-evident), 3= sufficient (sufficiently self-evident), 4= good (clearly self-evident), 5= excellent (extremely self-evident). All participants had conspicuity scores from one ureter. Difference in average index ureter conspicuity scores between NIR-F & WL across all timepoints was calculated for each participant. These were categorized based on if NIR-F score was at least 1, 2, 3 and 4 points higher.
Time Frame: WL and NIR-F: 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 450, 480 minutes
Population: mITT for all cohorts with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Participants: White Light +Near-infrared Fluorescence (Only WL) | All Participants: White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 94 | 94
Score on a scale
  30 minutes: number analyzed (Participants) | 83 | 82
  30 minutes | 2.8 (1.5) | 4.3 (1.1)
  60 minutes: number analyzed (Participants) | 74 | 73
  60 minutes | 2.7 (1.4) | 4.3 (1.1)
  90 minutes: number analyzed (Participants) | 55 | 55
  90 minutes | 2.4 (1.4) | 4.2 (1.1)
  120 minutes: number analyzed (Participants) | 40 | 40
  120 minutes | 2.4 (1.4) | 4.2 (1.1)
  150 minutes: number analyzed (Participants) | 27 | 27
  150 minutes | 2.0 (1.3) | 3.7 (1.4)
  180 minutes: number analyzed (Participants) | 19 | 19
  180 minutes | 2.3 (1.5) | 3.7 (1.3)
  210 minutes: number analyzed (Participants) | 10 | 10
  210 minutes | 2.2 (1.8) | 3.7 (1.7)
  240 minutes: number analyzed (Participants) | 3 | 3
  240 minutes | 4.3 (0.6) | 4.7 (0.6)
  270 minutes: number analyzed (Participants) | 4 | 4
  270 minutes | 3.8 (1.3) | 4.5 (1.0)
  300 minutes: number analyzed (Participants) | 2 | 2
  300 minutes | 3.5 (2.1) | 5.0 (0.0)
  330 minutes: number analyzed (Participants) | 1 | 1
  330 minutes | 2.0 (NA) — Only one participant was analyzed hence, SD is not evaluable | 4.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  450 minutes: number analyzed (Participants) | 2 | 1
  450 minutes | 3.0 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed | 1.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  480 minutes: number analyzed (Participants) | 2 | 2
  480 minutes | 2.0 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed | 4.0 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed
Statistical Analysis 1: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; POP with at least 1 Point Higher = 67.01 — Difference in average index ureter conspicuity scores between NIR-F & WL across all timepoints was calculated for each participant. These were categorized based on if NIR-F score was at least 1 point higher. POP meeting this criterion was estimated
Statistical Analysis 2: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; POP with at least 2 point higher = 40.4 — Difference in average index ureter conspicuity scores between NIR-F & WL across all timepoints was calculated for each participant. These were categorized based on if NIR-F score was at least 2 points higher. POP meeting this criterion was estimated
Statistical Analysis 3: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; POP with at least 3 point higher = 20.2 — Difference in average index ureter conspicuity scores between NIR-F & WL across all timepoints was calculated for each participant. These were categorized based on if NIR-F score was at least 3 points higher. POP meeting this criterion was estimated
Statistical Analysis 4: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); Test type: Superiority; POP with at least 4 point higher = 2.1 — Difference in average index ureter conspicuity scores between NIR-F & WL across all timepoints was calculated for each participant. These were categorized based on if NIR-F score was at least 4 points higher. POP meeting this criterion was estimated

15. Secondary Outcome: Blinded Independent Central Reviewer (BICR) Conspicuity Score Difference in Ureter Between WL and NIR-F at 30 Minutes (Adult (Normal/Mild): WL/NIR-F) and Concordance Correlation Coefficient (CCC) Between Investigator and BICR Reader
Description: BICR's conspicuity assessment of the ureter was scored individually for each illumination mode using a 5-Point Likert Scale ranging from 1 to 5 where 1= none (not self-evident), 2= poor (somewhat self-evident), 3= sufficient (sufficiently self-evident), 4= good (clearly self-evident), 5= excellent (extremely self-evident). All participants had conspicuity scores from one ureter. Concordance correlation coefficient (CCC) measures the agreement between investigator and BICR reader for the value difference between WL + NIR-F at 30 min timepoint. Results were reported for Reader 2, Reader 3 and Reader 4. Descriptive data for Investigator Conspicuity Score Difference in Ureter Between WL and NIR-F at 30 minutes is reported in Outcome measure #1.
Time Frame: 30 minutes post dose (+/- 15 minutes)
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 72 | 72
score on a scale
  READER 2 | 1.5 (0.9) | 3.4 (1.4)
  READER 3 | 2.1 (1.3) | 3.2 (1.3)
  READER 4 | 2.0 (1.1) | 4.3 (1.4)
Statistical Analysis 1: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; p < 0.001, paired t test; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [1.6 to 2.2], Standard Error of Mean 0.2 — Mean Difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint
Statistical Analysis 2: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); CCC between BICR and investigator (95% CI), Reader 2; Test type: Other — It quantifies the degree of concordance between two measurements; correlation coefficient = 0.221, 95% CI 2-sided [-0.011 to 0.431]
Statistical Analysis 3: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; p < 0.001, paired t test; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.8 to 1.5], Standard Error of Mean 0.2 — Mean Difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint
Statistical Analysis 4: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); CCC between BICR and investigator (95% CI), Reader 3; Test type: Other — It quantifies the degree of concordance between two measurements; correlation coefficient = 0.053, 95% CI 2-sided [-0.181 to 0.282]
Statistical Analysis 5: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; p < 0.001, paired t test; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [1.9 to 2.6], Standard Error of Mean 0.2 — Mean Difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint
Statistical Analysis 6: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); CCC between BICR and investigator (95% CI), Reader 4; Test type: Other — It quantifies the degree of concordance between two measurements; correlation coefficient = 0.260, 95% CI 2-sided [0.030 to 0.464]

16. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F an Average of All Timepoints [Adult (Normal/Mild): WL/NIR-F] and CCC Between Investigator and BICR Reader
Description: BICR's conspicuity assessment of the ureter was scored individually for each illumination mode using a 5-Point Likert Scale ranging from 1 to 5 where 1= none (not self-evident), 2= poor (somewhat self-evident), 3= sufficient (sufficiently self-evident), 4= good (clearly self-evident), 5= excellent (extremely self-evident). All participants had conspicuity scores from one ureter. CCC is concordance correlation coefficient, & it measures agreement between investigator and BICR reader for value difference between WL at 30-mintimepoint & average of all NIR-F time points. Result were reported for Reader 2, Reader 3 and Reader 4. Descriptive data for Investigator Conspicuity Score Difference in Ureter Between WL at 30 minutes and NIR-F an average of all timepoints is reported in Outcome measure #2.
Time Frame: WL: 30 minutes(+/- 15 minutes); NIR-F: 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 480 minutes
Population: ITT with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 72 | 72
score on a scale
  Reader 2, 30 minutes | 1.5 (0.9) | 3.4 (1.4)
  Reader 2, 60 minutes: number analyzed (Participants) | 0 | 45
  Reader 2, 60 minutes |  | 3.5 (1.3)
  Reader 2, 90 minutes: number analyzed (Participants) | 0 | 39
  Reader 2, 90 minutes |  | 3.2 (1.4)
  Reader 2, 120 minutes: number analyzed (Participants) | 0 | 29
  Reader 2, 120 minutes |  | 3.1 (1.4)
  Reader 2, 150 minutes: number analyzed (Participants) | 0 | 20
  Reader 2, 150 minutes |  | 3.3 (1.5)
  Reader 2, 180 minutes: number analyzed (Participants) | 0 | 15
  Reader 2, 180 minutes |  | 3.1 (1.4)
  Reader 2, 210 minutes: number analyzed (Participants) | 0 | 7
  Reader 2, 210 minutes |  | 3.4 (1.4)
  Reader 2, 240 minutes: number analyzed (Participants) | 0 | 1
  Reader 2, 240 minutes |  | 4.0 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 2, 270 minutes: number analyzed (Participants) | 0 | 4
  Reader 2, 270 minutes |  | 3.3 (2.1)
  Reader 2, 300 minutes: number analyzed (Participants) | 0 | 1
  Reader 2, 300 minutes |  | 4.0 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 2, 330 minutes: number analyzed (Participants) | 0 | 1
  Reader 2, 330 minutes |  | 3.0 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 2, 480 minutes: number analyzed (Participants) | 0 | 1
  Reader 2, 480 minutes |  | 1.0 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 3, 30 minutes | 2.1 (1.3) | 3.2 (1.3)
  Reader 3, 60 minutes: number analyzed (Participants) | 0 | 45
  Reader 3, 60 minutes |  | 3.5 (1.3)
  Reader 3, 90 minutes: number analyzed (Participants) | 0 | 39
  Reader 3, 90 minutes |  | 3.4 (1.3)
  Reader 3, 120 minutes: number analyzed (Participants) | 0 | 29
  Reader 3, 120 minutes |  | 3.4 (1.3)
  Reader 3, 150 minutes: number analyzed (Participants) | 0 | 20
  Reader 3, 150 minutes |  | 3.4 (1.3)
  Reader 3, 180 minutes: number analyzed (Participants) | 0 | 15
  Reader 3, 180 minutes |  | 3.5 (1.5)
  Reader 3, 210 minutes: number analyzed (Participants) | 0 | 7
  Reader 3, 210 minutes |  | 3.6 (1.4)
  Reader 3, 240 minutes: number analyzed (Participants) | 0 | 1
  Reader 3, 240 minutes |  | 5.0 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 3, 270 minutes: number analyzed (Participants) | 0 | 4
  Reader 3, 270 minutes |  | 3.8 (1.4)
  Reader 3, 300 minutes: number analyzed (Participants) | 0 | 1
  Reader 3, 300 minutes |  | 3.0 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 3, 330 minutes: number analyzed (Participants) | 0 | 1
  Reader 3, 330 minutes |  | 2 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 3, 480 minutes: number analyzed (Participants) | 0 | 1
  Reader 3, 480 minutes |  | 1 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 4, 30 minute | 2.0 (1.1) | 4.3 (1.1)
  Reader 4, 60 minute: number analyzed (Participants) | 0 | 45
  Reader 4, 60 minute |  | 4.4 (1.3)
  Reader 4, 90 minute: number analyzed (Participants) | 0 | 39
  Reader 4, 90 minute |  | 4.5 (1.0)
  Reader 4, 120 minute: number analyzed (Participants) | 0 | 29
  Reader 4, 120 minute |  | 4.4 (0.9)
  Reader 4, 150 minute: number analyzed (Participants) | 0 | 20
  Reader 4, 150 minute |  | 4.7 (0.7)
  Reader 4, 180 minute: number analyzed (Participants) | 0 | 15
  Reader 4, 180 minute |  | 4.3 (1.0)
  Reader 4, 210 minute: number analyzed (Participants) | 0 | 7
  Reader 4, 210 minute |  | 4.3 (1.1)
  Reader 4, 240 minute: number analyzed (Participants) | 0 | 1
  Reader 4, 240 minute |  | 5.0 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 4, 270 minute: number analyzed (Participants) | 0 | 4
  Reader 4, 270 minute |  | 4.0 (1.4)
  Reader 4, 300 minute: number analyzed (Participants) | 0 | 1
  Reader 4, 300 minute |  | 5.0 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 4, 330 minute: number analyzed (Participants) | 0 | 1
  Reader 4, 330 minute |  | 5.0 (NA) — Only one participant was analyzed hence SD was not evaluable
  Reader 4, 480 minute: number analyzed (Participants) | 0 | 1
  Reader 4, 480 minute |  | 2.0 (NA) — Only one participant was analyzed hence SD was not evaluable
Statistical Analysis 1: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; p < 0.001, Sign test; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [1.4 to 2.0], Standard Error of Mean 0.1 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); CCC between BICR and investigator (95% CI), Reader 2; Test type: Other — It quantifies the degree of concordance between two measurements; correlation coefficient = 0.219, 95% CI 2-sided [-0.013 to 0.429]
Statistical Analysis 3: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; p < 0.001, Sign test; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [0.8 to 1.4], Standard Error of Mean 0.2 — Mean Difference was calculated by averaging over the differences between NIR-F scores at each time point and the 30-min WL score of the index ureter(left or right) for eachparticipant
Statistical Analysis 4: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); CCC between BICR and investigator (95% CI), Reader 3; Test type: Other — It quantifies the degree of concordance between two measurements; correlation coefficient = 0.043, 95% CI 2-sided [-0.191 to 0.272]
Statistical Analysis 5: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; p < 0.001, Sign test; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [1.8 to 2.5], Standard Error of Mean 0.2 — [estimate comment as in outcome 16, analysis 3]
Statistical Analysis 6: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); CCC between BICR and investigator (95% CI), Reader 4; Test type: Other — It quantifies the degree of concordance between two measurements; correlation coefficient = 0.245, 95% CI 2-sided [0.014 to 0.451]

17. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F at End of Surgery [Adult (Normal/Mild): WL/NIR-F] and CCC Between Investigator and BICR Reader
Description: BICR's conspicuity assessment of the ureter was scored individually for each illumination mode using a 5-Point Likert Scale ranging from 1 to 5 where 1= none (not self-evident), 2= poor (somewhat self-evident), 3= sufficient (sufficiently self-evident), 4= good (clearly self-evident), 5= excellent (extremely self-evident). All participants had conspicuity scores from one ureter. CCC is concordance correlation coefficient, and it measures the agreement between investigator and BICR reader for the value difference between WL at 30-min timepoint and the end of surgery score under NIR-F. Results were reported for Reader 2, Reader 3 and Reader 4. Descriptive data for Investigator Conspicuity Score Difference in Ureter Between WL at 30 minutes and NIR-F at end of Surgery is reported in Outcome measure #3.
Time Frame: WL: 30 minute post dose (+/- 15 minutes); NIR-F: End of surgery (Day 1)
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 72 | 72
score on a scale
  READER 2, 30 minutes: number analyzed (Participants) | 72 | 0
  READER 2, 30 minutes | 1.5 (0.9) |
  READER 2 End of surgery (Day 1): number analyzed (Participants) | 0 | 72
  READER 2 End of surgery (Day 1) |  | 3.0 (1.4)
  READER 3, 30 minutes: number analyzed (Participants) | 72 | 0
  READER 3, 30 minutes | 2.1 (1.3) |
  READER 3, End of surgery (Day 1): number analyzed (Participants) | 0 | 72
  READER 3, End of surgery (Day 1) |  | 3.0 (1.4)
  READER 4, 30 minutes: number analyzed (Participants) | 72 | 0
  READER 4, 30 minutes | 2.0 (1.1) |
  READER 4, End of surgery (Day 1): number analyzed (Participants) | 0 | 72
  READER 4, End of surgery (Day 1) |  | 4.0 (1.5)
Statistical Analysis 1: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; p < 0.001, paired t test; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [1.1 to 1.8], Standard Error of Mean 0.2 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); CCC between BICR and investigator (95% CI), Reader 2; Test type: Other — It quantifies the degree of concordance between two measurements; correlation coefficient = 0.339, 95% CI 2-sided [0.116 to 0.529]
Statistical Analysis 3: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; p < 0.001, paired t test; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [0.6 to 1.3], Standard Error of Mean 0.2 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); CCC between BICR and investigator (95% CI), Reader 3; Test type: Other — It quantifies the degree of concordance between two measurements; correlation coefficient = 0.186, 95% CI 2-sided [-0.048 to 0.400]
Statistical Analysis 5: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; p < 0.001, paired t test; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [1.6 to 2.3], Standard Error of Mean 0.2 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); CCC between BICR and investigator (95% CI), Reader 4; Test type: Other — It quantifies the degree of concordance between two measurements; correlation coefficient = 0.297, 95% CI 2-sided [0.070 to 0.495]

18. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL and NIR-F at 30 Minutes [Adolescent (Normal/Mild): WL/NIR-F
Description: BICR's conspicuity assessment of the ureter was scored individually for each illumination mode using a 5-Point Likert Scale ranging from 1 to 5 where 1= none (not self-evident), 2= poor (somewhat self-evident), 3= sufficient (sufficiently self-evident), 4= good (clearly self-evident), 5= excellent (extremely self-evident). All participants had conspicuity scores from one ureter. Results were reported for Reader 2, Reader 3 and Reader 4.
Time Frame: 30 minutes post dose (+/- 15 minutes)
Population: mITT in adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 14 | 14
score on a scale
  Reader 2 | 2.1 (1.2) | 3.9 (1.3)
  Reader 3 | 2.9 (1.4) | 4.1 (1.0)
  Reader 4 | 3.4 (1.4) | 4.8 (0.6)
Statistical Analysis 1: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; Mean Difference (Final Values) = 1.8, Standard Error of Mean 0.4 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint
Statistical Analysis 2: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; Mean Difference (Final Values) = 1.2, Standard Error of Mean 0.4 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint
Statistical Analysis 3: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; Mean Difference (Final Values) = 1.4, Standard Error of Mean 0.3 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint

19. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F an Average of All Timepoints [Adolescent (Normal/Mild): WL/NIR-F]
Description: as for outcome 18
Time Frame: WL: 30 minutes(+/- 15 minutes); NIR-F: 30, 60, 90, 120, 150, 180, 210 minutes
Population: mITT in adolescents with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 14 | 14
score on a scale
  Reader 2: 30 minutes | 2.1 (1.2) | 3.9 (1.3)
  Reader 2: 60 minutes: number analyzed (Participants) | 0 | 10
  Reader 2: 60 minutes |  | 3.4 (1.2)
  Reader 2: 90 minutes: number analyzed (Participants) | 0 | 4
  Reader 2: 90 minutes |  | 3.8 (1.3)
  Reader 2: 120 minutes: number analyzed (Participants) | 0 | 1
  Reader 2: 120 minutes |  | 4.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 2: 150 minutes: number analyzed (Participants) | 0 | 1
  Reader 2: 150 minutes |  | 2.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 2: 180 minutes: number analyzed (Participants) | 0 | 1
  Reader 2: 180 minutes |  | 3 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 2: 210 minutes: number analyzed (Participants) | 0 | 1
  Reader 2: 210 minutes |  | 1 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 3: 30 minutes | 2.9 (1.4) | 4.1 (1.0)
  Reader 3: 60 minutes: number analyzed (Participants) | 0 | 10
  Reader 3: 60 minutes |  | 3.4 (1.0)
  Reader 3: 90 minutes: number analyzed (Participants) | 0 | 4
  Reader 3: 90 minutes |  | 3.8 (1.0)
  Reader 3: 120 minutes: number analyzed (Participants) | 0 | 1
  Reader 3: 120 minutes |  | 3.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 3: 150 minutes: number analyzed (Participants) | 0 | 1
  Reader 3: 150 minutes |  | 3.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 3: 180 minutes: number analyzed (Participants) | 0 | 1
  Reader 3: 180 minutes |  | 3.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 3: 210 minutes: number analyzed (Participants) | 0 | 1
  Reader 3: 210 minutes |  | 1.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 4: 30 minutes | 3.4 (1.3) | 4.8 (0.6)
  Reader 4: 60 minutes: number analyzed (Participants) | 0 | 10
  Reader 4: 60 minutes |  | 5.0 (0.0)
  Reader 4: 90 minutes: number analyzed (Participants) | 0 | 4
  Reader 4: 90 minutes |  | 5.0 (0.0)
  Reader 4: 120 minutes: number analyzed (Participants) | 0 | 1
  Reader 4: 120 minutes |  | 5.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 4: 150 minutes: number analyzed (Participants) | 0 | 1
  Reader 4: 150 minutes |  | 5.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 4: 180 minutes: number analyzed (Participants) | 0 | 1
  Reader 4: 180 minutes |  | 5.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 4: 210 minutes: number analyzed (Participants) | 0 | 1
  Reader 4: 210 minutes |  | 5.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
Statistical Analysis 1: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); Difference from WL in Means, Reader 2; Test type: Superiority; Mean Difference (Final Values) = 1.5, Standard Error of Mean 0.3 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); Difference from WL in Means, Reader 3; Test type: Superiority; Mean Difference (Final Values) = 0.9, Standard Error of Mean 0.4 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); Difference from WL in Means, Reader 4; Test type: Superiority; Mean Difference (Final Values) = 1.5, Standard Error of Mean 0.3 — [estimate comment as in outcome 6, analysis 1]

20. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F at End of Surgery [Adolescent (Normal/Mild): WL/NIR-F]
Description: as for outcome 18
Time Frame: WL: 30 minute post dose (+/- 15 minutes); NIR-F: End of surgery (Day 1)
Population: mITT in adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) | Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 14 | 14
score on a scale
  Reader 2: 30 minutes: number analyzed (Participants) | 14 | 0
  Reader 2: 30 minutes | 2.1 (1.2) |
  Reader 2: End of surgery (Day 1): number analyzed (Participants) | 0 | 14
  Reader 2: End of surgery (Day 1) |  | 3.4 (1.5)
  Reader 3: 30 minutes: number analyzed (Participants) | 14 | 0
  Reader 3: 30 minutes | 2.9 (1.4) |
  Reader 3: End of surgery (Day 1): number analyzed (Participants) | 0 | 14
  Reader 3: End of surgery (Day 1) |  | 3.6 (1.3)
  Reader 4: 30 minutes: number analyzed (Participants) | 14 | 0
  Reader 4: 30 minutes | 3.4 (1.3) |
  Reader 4: End of surgery (Day 1): number analyzed (Participants) | 0 | 14
  Reader 4: End of surgery (Day 1) |  | 4.8 (0.6)
Statistical Analysis 1: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; Mean Difference (Final Values) = 1.2, Standard Error of Mean 0.4 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; Mean Difference (Final Values) = 0.7, Standard Error of Mean 0.4 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only WL) vs Adolescent (Normal/Mild): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; Mean Difference (Final Values) = 1.4, Standard Error of Mean 0.3 — [estimate comment as in outcome 3, analysis 1]

21. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL and NIR-F at 30 Minutes [Adult (Moderate): WL/NIR-F]
Description: as for outcome 18
Time Frame: 30 minutes post dose (+/- 15 minutes)
Population: mITT in adults with moderate eGFR
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) | Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 8 | 8
score on a scale
  Reader 2 | 1.3 (0.7) | 2.4 (1.4)
  Reader 3 | 1.5 (0.5) | 2.4 (1.1)
  Reader 4 | 2.0 (0.9) | 4.1 (1.4)
Statistical Analysis 1: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; Mean Difference (Final Values) = 1.1, Standard Error of Mean 0.4 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint
Statistical Analysis 2: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; Mean Difference (Final Values) = 0.9, Standard Error of Mean 0.3 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint
Statistical Analysis 3: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; Mean Difference (Final Values) = 2.1, Standard Error of Mean 0.5 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint

22. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F an Average of All Timepoints [Adult (Moderate): WL/NIR-F]
Description: as for outcome 18
Time Frame: WL: 30 minutes(+/- 15 minutes); NIR-F: 30, 60, 90, 120, 150, 180 minutes
Population: mITT in adults with moderate eGFR with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) | Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 8 | 8
score on a scale
  Reader 2: 30 minutes | 1.3 (0.7) | 2.4 (1.4)
  Reader 2: 60 minutes: number analyzed (Participants) | 0 | 2
  Reader 2: 60 minutes |  | 3.5 (2.1)
  Reader 2: 90 minutes: number analyzed (Participants) | 0 | 4
  Reader 2: 90 minutes |  | 2.8 (1.5)
  Reader 2: 120 minutes: number analyzed (Participants) | 0 | 4
  Reader 2: 120 minutes |  | 2.8 (1.7)
  Reader 2: 150 minutes: number analyzed (Participants) | 0 | 3
  Reader 2: 150 minutes |  | 2.3 (0.6)
  Reader 2: 180 minutes: number analyzed (Participants) | 0 | 1
  Reader 2: 180 minutes |  | 1 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 3: 30 minutes | 1.5 (0.5) | 2.4 (1.1)
  Reader 3: 60 minutes: number analyzed (Participants) | 0 | 2
  Reader 3: 60 minutes |  | 3.5 (2.1)
  Reader 3: 90 minutes: number analyzed (Participants) | 0 | 4
  Reader 3: 90 minutes |  | 2.8 (1.5)
  Reader 3: 120 minutes: number analyzed (Participants) | 0 | 4
  Reader 3: 120 minutes |  | 3.0 (1.6)
  Reader 3: 150 minutes: number analyzed (Participants) | 0 | 3
  Reader 3: 150 minutes |  | 2.3 (0.6)
  Reader 3: 180 minutes: number analyzed (Participants) | 0 | 1
  Reader 3: 180 minutes |  | 2.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 4: 30 minutes | 2.0 (0.9) | 4.1 (1.4)
  Reader 4: 60 minutes: number analyzed (Participants) | 0 | 2
  Reader 4: 60 minutes |  | 4.5 (0.7)
  Reader 4: 90 minutes: number analyzed (Participants) | 0 | 4
  Reader 4: 90 minutes |  | 5.0 (0.0)
  Reader 4: 120 minutes: number analyzed (Participants) | 0 | 4
  Reader 4: 120 minutes |  | 3.8 (1.5)
  Reader 4: 150 minutes: number analyzed (Participants) | 0 | 3
  Reader 4: 150 minutes |  | 4.7 (0.6)
  Reader 4: 180 minutes: number analyzed (Participants) | 0 | 1
  Reader 4: 180 minutes |  | 4.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
Statistical Analysis 1: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; Mean Difference (Final Values) = 1.1, Standard Error of Mean 0.3 — Mean Difference was calculated by averaging over the differences between NIR-F scores at each time point and the 30-m in WL score of the ureter of interest (left; right) for each participant
Statistical Analysis 2: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; Mean Difference (Final Values) = 1.1, Standard Error of Mean 0.3 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; Mean Difference (Final Values) = 1.0, Standard Error of Mean 0.3 — [estimate comment as in outcome 6, analysis 1]

23. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F at End of Surgery [Adult (Moderate): WL/NIR-F]
Description: as for outcome 18
Time Frame: WL: 30 minute post dose (+/- 15 minutes); NIR-F: End of surgery (Day 1)
Population: mITT in adults with moderate eGFR
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) | Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 8 | 8
score on a scale
  Reader 2: 30 minutes: number analyzed (Participants) | 8 | 0
  Reader 2: 30 minutes | 1.3 (0.7) |
  Reader 2: End of Surgery (Day 1): number analyzed (Participants) | 0 | 8
  Reader 2: End of Surgery (Day 1) |  | 2.3 (1.3)
  Reader 3: 30 minutes: number analyzed (Participants) | 8 | 0
  Reader 3: 30 minutes | 1.5 (0.5) |
  Reader 3: End of Surgery (Day 1): number analyzed (Participants) | 0 | 8
  Reader 3: End of Surgery (Day 1) |  | 2.6 (1.1)
  Reader 4: 30 minutes: number analyzed (Participants) | 8 | 0
  Reader 4: 30 minutes | 2.0 (0.9) |
  Reader 4: End of Surgery (Day 1): number analyzed (Participants) | 0 | 8
  Reader 4: End of Surgery (Day 1) |  | 4.0 (1.1)
Statistical Analysis 1: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; Mean Difference (Final Values) = 1.0, Standard Error of Mean 0.3 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; Mean Difference (Final Values) = 1.1, Standard Error of Mean 0.4 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Adult (Moderate): White Light +Near-infrared Fluorescence (Only WL) vs Adult (Moderate): White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; Mean Difference (Final Values) = 2.0, Standard Error of Mean 0.5 — [estimate comment as in outcome 3, analysis 1]

24. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL and NIR-F at 30 Minutes [All Participants]
Description: as for outcome 18
Time Frame: 30 minutes post dose (+/- 15 minutes)
Population: mITT for all cohorts in WL/NIR-F arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants: White Light +Near-infrared Fluorescence (Only WL) | All Participants: White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 94 | 94
score on a scale
  Reader 2 | 1.6 (0.9) | 3.4 (1.4)
  Reader 3 | 2.1 (1.3) | 3.3 (1.3)
  Reader 4 | 2.2 (1.2) | 4.4 (1.3)
Statistical Analysis 1: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; Mean Difference (Final Values) = 1.8, Standard Error of Mean 0.1 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint
Statistical Analysis 2: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; Mean Difference (Final Values) = 1.1, Standard Error of Mean 0.1 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint
Statistical Analysis 3: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; Mean Difference (Final Values) = 2.1, Standard Error of Mean 0.1 — Mean difference was calculated by averaging over the differences between WL scores and NIR-F scores at 30-min timepoint

25. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F an Average of All Timepoints [All Participants]
Description: as for outcome 18
Time Frame: WL: 30 minutes(+/- 15 minutes); NIR-F: 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 480 minutes
Population: mITT for all cohorts in WL/NIR-F arm with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants: White Light +Near-infrared Fluorescence (Only WL) | All Participants: White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 94 | 94
score on a scale
  Reader 2: 30 minutes | 1.6 (0.9) | 3.4 (1.4)
  Reader 2: 60 minutes: number analyzed (Participants) | 0 | 57
  Reader 2: 60 minutes |  | 3.5 (1.3)
  Reader 2: 90 minutes: number analyzed (Participants) | 0 | 47
  Reader 2: 90 minutes |  | 3.2 (1.4)
  Reader 2: 120 minutes: number analyzed (Participants) | 0 | 34
  Reader 2: 120 minutes |  | 3.1 (1.4)
  Reader 2: 150 minutes: number analyzed (Participants) | 0 | 24
  Reader 2: 150 minutes |  | 3.1 (1.4)
  Reader 2: 180 minutes: number analyzed (Participants) | 0 | 17
  Reader 2: 180 minutes |  | 3.0 (1.4)
  Reader 2: 210 minutes: number analyzed (Participants) | 0 | 8
  Reader 2: 210 minutes |  | 3.1 (1.6)
  Reader 2: 240 minutes: number analyzed (Participants) | 0 | 1
  Reader 2: 240 minutes |  | 4.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 2: 270 minutes: number analyzed (Participants) | 0 | 4
  Reader 2: 270 minutes |  | 3.3 (2.1)
  Reader 2: 300 minutes: number analyzed (Participants) | 0 | 1
  Reader 2: 300 minutes |  | 4.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 2: 330 minutes: number analyzed (Participants) | 0 | 1
  Reader 2: 330 minutes |  | 3.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 2: 480 minutes: number analyzed (Participants) | 0 | 1
  Reader 2: 480 minutes |  | 1.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 3: 30 minutes | 2.1 (1.3) | 3.3 (1.3)
  Reader 3: 60 minutes: number analyzed (Participants) | 0 | 57
  Reader 3: 60 minutes |  | 3.5 (1.2)
  Reader 3: 90 minutes: number analyzed (Participants) | 0 | 47
  Reader 3: 90 minutes |  | 3.4 (1.3)
  Reader 3: 120 minutes: number analyzed (Participants) | 0 | 34
  Reader 3: 120 minutes |  | 3.3 (1.3)
  Reader 3: 150 minutes: number analyzed (Participants) | 0 | 24
  Reader 3: 150 minutes |  | 3.3 (1.4)
  Reader 3: 180 minutes: number analyzed (Participants) | 0 | 17
  Reader 3: 180 minutes |  | 3.4 (1.4)
  Reader 3: 210 minutes: number analyzed (Participants) | 0 | 8
  Reader 3: 210 minutes |  | 3.3 (1.6)
  Reader 3: 240 minutes: number analyzed (Participants) | 0 | 1
  Reader 3: 240 minutes |  | 5.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 3: 270 minutes: number analyzed (Participants) | 0 | 4
  Reader 3: 270 minutes |  | 3.8 (1.9)
  Reader 3: 300 minutes: number analyzed (Participants) | 0 | 1
  Reader 3: 300 minutes |  | 3.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 3: 330 minutes: number analyzed (Participants) | 0 | 1
  Reader 3: 330 minutes |  | 2.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 3: 480 minutes: number analyzed (Participants) | 0 | 1
  Reader 3: 480 minutes |  | 1.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 4: 30 minutes | 2.2 (1.2) | 4.4 (1.3)
  Reader 4: 60 minutes: number analyzed (Participants) | 0 | 57
  Reader 4: 60 minutes |  | 4.5 (1.2)
  Reader 4: 90 minutes: number analyzed (Participants) | 0 | 47
  Reader 4: 90 minutes |  | 4.6 (0.9)
  Reader 4:120 minutes: number analyzed (Participants) | 0 | 34
  Reader 4:120 minutes |  | 4.4 (1.0)
  Reader 4: 150 minutes: number analyzed (Participants) | 0 | 24
  Reader 4: 150 minutes |  | 4.7 (0.7)
  Reader 4: 180 minutes: number analyzed (Participants) | 0 | 17
  Reader 4: 180 minutes |  | 4.3 (1.0)
  Reader 4: 210 minutes: number analyzed (Participants) | 0 | 8
  Reader 4: 210 minutes |  | 4.1 (1.1)
  Reader 4: 240 minutes: number analyzed (Participants) | 0 | 1
  Reader 4: 240 minutes |  | 5.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 4: 270 minutes: number analyzed (Participants) | 0 | 4
  Reader 4: 270 minutes |  | 4.0 (1.4)
  Reader 4: 300 minutes: number analyzed (Participants) | 0 | 1
  Reader 4: 300 minutes |  | 5.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 4: 330 minutes: number analyzed (Participants) | 0 | 1
  Reader 4: 330 minutes |  | 5.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
  Reader 4: 480 minutes: number analyzed (Participants) | 0 | 1
  Reader 4: 480 minutes |  | 2.0 (NA) — Only one participant was analyzed hence, SD is not evaluable
Statistical Analysis 1: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; Mean Difference (Final Values) = 1.6, Standard Error of Mean 0.1 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; Mean Difference (Final Values) = 1.1, Standard Error of Mean 0.1 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; Mean Difference (Final Values) = 2.1, Standard Error of Mean 0.1 — [estimate comment as in outcome 6, analysis 1]

26. Secondary Outcome: BICR Conspicuity Score Difference in Ureter Between WL at 30 Minutes and NIR-F at End of Surgery [All Participants]
Description: as for outcome 18
Time Frame: WL: 30 minute post dose (+/- 15 minutes); NIR-F: End of surgery (Day 1)
Population: mITT for all cohorts in WL/NIR-F arm
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: White Light +Near-infrared Fluorescence (Only NIR-F): Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult and adolescent participants with normal renal function or mild or moderate renal impairment. WL and NIR-F were used to recognize/identify the ureter. Only NIRF was reported for this arm.
Arm/Group | All Participants: White Light +Near-infrared Fluorescence (Only WL) | All Participants: White Light +Near-infrared Fluorescence (Only NIR-F)
Number analyzed (Participants) | 94 | 94
score on a scale
  Reader 2: 30 minutes: number analyzed (Participants) | 94 | 0
  Reader 2: 30 minutes | 1.6 (0.9) |
  Reader 2: End of surgery (Day 1): number analyzed (Participants) | 0 | 94
  Reader 2: End of surgery (Day 1) |  | 3.0 (1.4)
  Reader 3: 30 minutes: number analyzed (Participants) | 94 | 0
  Reader 3: 30 minutes | 2.1 (1.3) |
  Reader 3: End of surgery (Day 1): number analyzed (Participants) | 0 | 94
  Reader 3: End of surgery (Day 1) |  | 3.1 (1.4)
  Reader 4: 30 minutes: number analyzed (Participants) | 94 | 0
  Reader 4: 30 minutes | 2.2 (1.2) |
  Reader 4: End of surgery (Day 1): number analyzed (Participants) | 0 | 94
  Reader 4: End of surgery (Day 1) |  | 4.1 (1.4)
Statistical Analysis 1: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); For reader 2; Test type: Superiority; Mean Difference (Final Values) = 1.4, Standard Error of Mean 0.2 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); For reader 3; Test type: Superiority; Mean Difference (Final Values) = 0.9, Standard Error of Mean 0.2 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: All Participants: White Light +Near-infrared Fluorescence (Only WL) vs All Participants: White Light +Near-infrared Fluorescence (Only NIR-F); For reader 4; Test type: Superiority; Mean Difference (Final Values) = 1.9, Standard Error of Mean 0.2 — [estimate comment as in outcome 3, analysis 1]

27. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered an Investigational Product (IP) and which does not necessarily had a causal relationship with the treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding; abnormal laboratory test result or other safety assessment, symptom, or disease temporally associated with the use of IP whether considered related to the IP. A TEAE was defined as an AE with onset at any time from first dosing until the follow up period. AEs were considered serious (SAEs) if the AE resulted, in death, was life-threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly, or birth defect or required inpatient hospitalization or led to prolongation of hospitalization. TEAEs included both serious and Other (Not Including Serious) TEAE.
Time Frame: From first dose up to 15 days (+ 10 days)
Population: SAF
Measure: Number; unit: participants
Groups:
- Adult (Moderate): White Light/ Near-infrared Fluorescence: Pudexacianinium (3mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adult participants with moderate renal impairment. WL and NIR-F were used to recognize/identify the ureter.
- Adolescent (Normal/Mild): White Light/ Near-infrared Fluorescence: Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 min before ureter visualization, on Day 1 in adolescent participants with normal renal function or mild renal impairment. WL and NIR-F were used to recognize/identify the ureter.
Arm/Group | Adult (Normal/Mild): White Light Only | Adult (Normal/Mild): White Light/Near-infrared Fluorescence | Adult (Moderate): White Light/ Near-infrared Fluorescence | Adolescent (Normal/Mild): White Light/ Near-infrared Fluorescence
Number analyzed (Participants) | 13 | 70 | 8 | 14
participants
  TEAE | 8 | 28 | 1 | 7
  Serious TEAE | 4 | 8 | 0 | 0

28. Secondary Outcome: Pharmacokinetics (PK) of Pudexacianinium Chloride: Plasma Concentration
Description: Concentration of pudexacianinium chloride in plasma. PK samples were collected up to the end of surgery timepoint of each participant. As planned SD was reported only if >=3 participants were evaluated for a specific timepoint.
Time Frame: Day 1 Postdose: 10, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 390, 360 minutes
Population: Pharmacokinetic Analysis Set (PKAS): All participants in any cohort who received pudexacianinium chloride for which at least 1 plasma or urine concentration data was available with the time for dosing and sampling. Since participants had different end of surgery timepoint, number of observations were different by Arm/Group as the last observation timepoint is different by participant. PKAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: nanogram/milliliters (ng/mL)
Groups:
- Adult (Normal/Mild): White Light/ Near-infrared Fluorescence: Pudexacianinium (3 mg) was administered as a single IV dose approximately 30 minutes min before ureter visualization, on Day 1 in adult participants with normal renal function or mild renal impairment. WL and NIR-F were used to recognize/identify the ureter.
Arm/Group | Adult (Normal/Mild): White Light Only | Adult (Normal/Mild): White Light/ Near-infrared Fluorescence | Adult (Moderate): White Light/ Near-infrared Fluorescence | Adolescent (Normal/Mild): White Light/ Near-infrared Fluorescence
Number analyzed (Participants) | 13 | 62 | 8 | 14
nanogram/milliliters (ng/mL)
  10 minutes | 366 (109) | 411 (387) | 426 (137) | 410 (141)
  30 minutes: number analyzed (Participants) | 13 | 61 | 8 | 14
  30 minutes | 197 (61.2) | 185 (46.8) | 267 (93.6) | 244 (86.4)
  60 minutes: number analyzed (Participants) | 11 | 59 | 8 | 12
  60 minutes | 129 (34.4) | 126 (36.1) | 203 (56.8) | 166 (50.1)
  90 minutes: number analyzed (Participants) | 7 | 30 | 5 | 9
  90 minutes | 111 (40.5) | 108 (34.6) | 172 (42.3) | 121 (46.1)
  120 minutes: number analyzed (Participants) | 8 | 45 | 6 | 8
  120 minutes | 78.3 (37.1) | 79.8 (30.3) | 147 (44.7) | 99.2 (26.8)
  150 minutes: number analyzed (Participants) | 3 | 21 | 4 | 2
  150 minutes | 115 (37.3) | 82.8 (29.0) | 128 (25.1) | 120 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed
  180 minutes: number analyzed (Participants) | 6 | 20 | 2 | 3
  180 minutes | 59.2 (24.1) | 61.9 (24.8) | 128 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed | 47.1 (17.5)
  210 minutes: number analyzed (Participants) | 2 | 5 | 1 | 0
  210 minutes | 47.8 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed | 53.8 (16.0) | 97.6 (NA) — Only one participant was analyzed, hence SD is not evaluable |
  240 minutes: number analyzed (Participants) | 1 | 5 | 0 | 0
  240 minutes | 45.8 (NA) — Only 1 participant was analyzed, hence SD was not evaluable. | 69.7 (28.5) |  |
  270 minutes: number analyzed (Participants) | 0 | 2 | 0 | 1
  270 minutes |  | 42.4 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  | 34.2 (NA) — Only one participant was analyzed, hence SD was not evaluable
  300 minutes: number analyzed (Participants) | 1 | 3 | 0 | 0
  300 minutes | 30.9 (NA) — Only one participant was analyzed hence, SD is not evaluable | 51.1 (18.7) |  |
  330 minutes: number analyzed (Participants) | 0 | 1 | 0 | 0
  330 minutes |  | 25.6 (NA) — Only one participant was analyzed hence, SD is not evaluable |  |
  360 minutes: number analyzed (Participants) | 0 | 1 | 0 | 0
  360 minutes |  | 22.4 (NA) — Only one participant was analyzed hence, SD is not evaluable |  |
  390 minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  390 minutes |  | 28.9 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  |

29. Secondary Outcome: PK of Pudexacianinium Chloride: Urine Concentration
Description: Concentration of pudexacianinium chloride in urine.PK samples were collected up to the end of surgery timepoint of each participant. PK samples were collected up to the end of surgery timepoint of each participant. As planned SD was reported only if >=3 participants were evaluated for a specific timepoint.
Time Frame: Day 1 Postdose: 0-10, 10-30, 30-60, 60-90, 90-120, 120-150, 150-180, 180-210, 210-240, 240-270, 270-300, 300-330, 330-360, 360-390, 390-420, 420-450, 450-480 minutes
Population: PKAS with available data was analyzed. Since participants had different end of surgery timepoint, number of observations were different by Arm/Group as the last observation timepoint is different by participant.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Adult (Normal/Mild): White Light Only | Adult (Normal/Mild): White Light/ Near-infrared Fluorescence | Adult (Moderate): White Light/ Near-infrared Fluorescence | Adolescent (Normal/Mild): White Light/ Near-infrared Fluorescence
Number analyzed (Participants) | 11 | 56 | 8 | 13
ng/mL
  0-10 minutes: number analyzed (Participants) | 11 | 56 | 8 | 9
  0-10 minutes | 1530 (4100) | 235 (629) | 80.4 (165) | 9.98 (29.9)
  10-30 minutes: number analyzed (Participants) | 10 | 51 | 4 | 13
  10-30 minutes | 4960 (6050) | 10200 (15600) | 7890 (3610) | 14200 (15100)
  30-60 minutes: number analyzed (Participants) | 9 | 52 | 3 | 13
  30-60 minutes | 18000 (18600) | 19800 (20300) | 10400 (6640) | 25200 (22000)
  60-90 minutes: number analyzed (Participants) | 8 | 47 | 6 | 7
  60-90 minutes | 16700 (18100) | 20100 (21200) | 25500 (17100) | 41600 (41900)
  90-120 minutes: number analyzed (Participants) | 5 | 35 | 5 | 5
  90-120 minutes | 17700 (13300) | 14500 (9630) | 25800 (37200) | 49800 (62000)
  120-150 minutes: number analyzed (Participants) | 5 | 24 | 2 | 5
  120-150 minutes | 20700 (8850) | 10700 (6880) | 17400 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed | 25500 (16600)
  150-180 minutes: number analyzed (Participants) | 5 | 22 | 1 | 2
  150-180 minutes | 17900 (7900) | 9110 (6530) | 18400 (NA) — Only one participant was analyzed hence, SD is not evaluable | 19600 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed
  180-210 minutes: number analyzed (Participants) | 1 | 5 | 0 | 1
  180-210 minutes | 6230 (NA) — Only one participant was analyzed hence, SD is not evaluable | 8690 (6920) |  | 10500 (NA) — Only one participant was analyzed hence, SD is not evaluable
  210-240 minutes: number analyzed (Participants) | 1 | 4 | 0 | 1
  210-240 minutes | 5230 (NA) — Only one participant was analyzed hence, SD is not evaluable | 5750 (2310) |  | 6500 (NA) — Only one participant was analyzed hence, SD is not evaluable
  240-270 minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  240-270 minutes |  | 5500 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  |
  270- 300 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  270- 300 minutes |  | 3690 (1600) |  |
  300- 330 minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  300- 330 minutes |  | 4860 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  |
  330- 360 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  330- 360 minutes |  | 3630 (2280) |  |
  360-390 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  360-390 minutes |  | 2650 (1640) |  |
  390-420 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  390-420 minutes |  | 1570 (2400) |  |
  420-450 minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  420-450 minutes |  | 3150 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  |
  450-480 minutes: number analyzed (Participants) | 0 | 1 | 0 | 0
  450-480 minutes |  | 3070 (NA) — Only one participant was analyzed hence, SD is not evaluable |  |

30. Secondary Outcome: Amount of Pudexacianinium Chloride Excreted Into Urine (Ae)
Description: PK samples were collected up to the end of surgery timepoint of each participant. As planned SD was reported only if >=3 participants were evaluated for a specific timepoint.
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Adult (Normal/Mild): White Light Only | Adult (Normal/Mild): White Light/ Near-infrared Fluorescence | Adult (Moderate): White Light/ Near-infrared Fluorescence | Adolescent (Normal/Mild): White Light/ Near-infrared Fluorescence
Number analyzed (Participants) | 10 | 56 | 8 | 13
milligrams
  0-10 minutes: number analyzed (Participants) | 10 | 56 | 8 | 9
  0-10 minutes | 0.0443 (0.0790) | 0.0190 (0.0425) | 0.00713 (0.0194) | 0.000657 (0.00197)
  10-30 minutes: number analyzed (Participants) | 9 | 51 | 4 | 13
  10-30 minutes | 0.0773 (0.122) | 0.164 (0.198) | 0.122 (0.0759) | 0.245 (0.269)
  30-60 minutes: number analyzed (Participants) | 9 | 52 | 3 | 13
  30-60 minutes | 0.375 (0.276) | 0.274 (0.230) | 0.175 (0.0305) | 0.240 (0.258)
  60-90 minutes: number analyzed (Participants) | 8 | 48 | 6 | 7
  60-90 minutes | 0.304 (0.290) | 0.340 (0.232) | 0.216 (0.160) | 0.348 (0.417)
  90-120 minutes: number analyzed (Participants) | 5 | 36 | 5 | 5
  90-120 minutes | 0.325 (0.261) | 0.306 (0.199) | 0.151 (0.0570) | 0.578 (0.465)
  120-150 minutes: number analyzed (Participants) | 5 | 24 | 2 | 5
  120-150 minutes | 0.301 (0.112) | 0.203 (0.131) | 0.0511 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed | 0.256 (0.170)
  150-180 minutes: number analyzed (Participants) | 5 | 22 | 1 | 2
  150-180 minutes | 0.286 (0.289) | 0.143 (0.0859) | 0.171 (NA) — Only one participant was analyzed hence, SD is not evaluable | 0.450 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed
  180-210 minutes: number analyzed (Participants) | 1 | 5 | 0 | 1
  180-210 minutes | 0.147 (NA) — Only one participant was analyzed hence, SD is not evaluable | 0.151 (0.0763) |  | 0.162 (NA) — Only one participant was analyzed hence, SD is not evaluable
  210-240 minutes: number analyzed (Participants) | 1 | 4 | 0 | 1
  210-240 minutes | 0.175 (NA) — Only one participant was analyzed hence, SD is not evaluable | 0.0937 (0.0307) |  | 0.0702 (NA) — Only one participant was analyzed hence, SD is not evaluable
  240-270 minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  240-270 minutes |  | 0.0803 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  |
  270- 300 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  270- 300 minutes |  | 0.0655 (0.0105) |  |
  300- 330 minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  300- 330 minutes |  | 0.0582 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  |
  330- 360 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  330- 360 minutes |  | 0.0438 (0.0541) |  |
  360-390 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  360-390 minutes |  | 0.0808 (0.0412) |  |
  390-420 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  390-420 minutes |  | 0.0263 (0.0209) |  |
  420-450 minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  420-450 minutes |  | 0.0835 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  |
  450- 480 minutes: number analyzed (Participants) | 0 | 1 | 0 | 0
  450- 480 minutes |  | 0.0301 (NA) — Only one participant was analyzed hence, SD is not evaluable |  |

31. Secondary Outcome: Percentage of Pudexacianinium Chloride Dose Excreted Into Urine (Ae%)
Description: as for outcome 30
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: percentage of drug excreted
Arm/Group | Adult (Normal/Mild): White Light Only | Adult (Normal/Mild): White Light/ Near-infrared Fluorescence | Adult (Moderate): White Light/ Near-infrared Fluorescence | Adolescent (Normal/Mild): White Light/ Near-infrared Fluorescence
Number analyzed (Participants) | 10 | 56 | 8 | 13
percentage of drug excreted
  0-10 minutes: number analyzed (Participants) | 10 | 56 | 8 | 9
  0-10 minutes | 1.48 (2.63) | 0.633 (1.42) | 0.238 (0.646) | 0.0219 (0.0657)
  10-30 minutes: number analyzed (Participants) | 9 | 51 | 4 | 13
  10-30 minutes | 2.58 (4.06) | 5.46 (6.59) | 4.06 (2.53) | 8.18 (8.98)
  30-60 minutes: number analyzed (Participants) | 9 | 52 | 3 | 13
  30-60 minutes | 12.5 (9.21) | 9.15 (7.68) | 5.83 (1.02) | 7.99 (8.59)
  60-90 minutes: number analyzed (Participants) | 8 | 48 | 6 | 7
  60-90 minutes | 10.1 (9.66) | 11.3 (7.74) | 7.20 (5.32) | 11.6 (13.9)
  90-120 minutes: number analyzed (Participants) | 5 | 36 | 5 | 5
  90-120 minutes | 10.8 (8.71) | 10.2 (6.63) | 5.03 (1.90) | 19.3 (15.5)
  120-150 minutes: number analyzed (Participants) | 5 | 24 | 2 | 5
  120-150 minutes | 10.0 (3.74) | 6.77 (4.38) | 1.70 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed | 8.54 (5.68)
  150-180 minutes: number analyzed (Participants) | 5 | 22 | 1 | 2
  150-180 minutes | 9.52 (9.62) | 4.78 (2.86) | 5.70 (NA) — Only one participant was analyzed, hence SD was not evaluable | 15.0 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed
  180-210 minutes: number analyzed (Participants) | 1 | 5 | 0 | 1
  180-210 minutes | 4.90 (NA) — Only one participant was analyzed, hence SD was not evaluable | 5.03 (2.54) |  | 5.39 (NA) — Only one participant was analyzed, hence SD was not evaluable
  210-240 minutes: number analyzed (Participants) | 1 | 4 | 0 | 1
  210-240 minutes | 5.82 (NA) — Only one participant was analyzed, hence SD was not evaluable | 3.12 (1.02) |  | 2.34 (NA) — Only one participant was analyzed, hence SD was not evaluable
  240-270 minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  240-270 minutes |  | 2.68 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  |
  270- 300 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  270- 300 minutes |  | 2.18 (0.351) |  |
  300- 330 minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  300- 330 minutes |  | 1.94 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  |
  330- 360 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  330- 360 minutes |  | 1.46 (1.80) |  |
  360-390 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  360-390 minutes |  | 2.69 (1.37) |  |
  390-420 minutes: number analyzed (Participants) | 0 | 3 | 0 | 0
  390-420 minutes |  | 0.877 (0.697) |  |
  420-450 minutes: number analyzed (Participants) | 0 | 2 | 0 | 0
  420-450 minutes |  | 2.78 (NA) — Based on an internal programming guideline SD was reported if at least 3 participants were analyzed |  |
  450-480 minutes: number analyzed (Participants) | 0 | 1 | 0 | 0
  450-480 minutes |  | 1.00 (NA) — Only one participant was analyzed, hence SD was not evaluable |  |

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM): From randomization up to 15 days (+ 10 days) AE- From first dose up to 15 days (+ 10 days)
Description: Participants at risk in ACM was collected and analyzed for all enrolled/randomized population. Participants at risk in Serious and Non serious adverse events were collected and analyzed in the SAF (dosed with ASP5354).
Arm/Group | Adult (Normal/Mild): White Light/Near-infrared Fluorescence | Adult (Normal/Mild): White Light Only | Adult (Moderate): White Light/Near-infrared Fluorescence | Adolescent (Normal/Mild): WL/NIR-F
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/13 | 0/8 | 0/14
Serious Adverse Events (participants affected / at risk) | 8/70 | 4/13 | 0/8 | 0/14
Other Adverse Events (participants affected / at risk) | 11/70 | 5/13 | 1/8 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult (Normal/Mild): White Light/Near-infrared Fluorescence (N=70) | Adult (Normal/Mild): White Light Only (N=13) | Adult (Moderate): White Light/Near-infrared Fluorescence (N=8) | Adolescent (Normal/Mild): WL/NIR-F (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult (Normal/Mild): White Light/Near-infrared Fluorescence (N=70) | Adult (Normal/Mild): White Light Only (N=13) | Adult (Moderate): White Light/Near-infrared Fluorescence (N=8) | Adolescent (Normal/Mild): WL/NIR-F (N=14)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dilutional anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Loss of bladder sensation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT05754333/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT05754333/SAP_001.pdf